CLINICAL TRIAL: NCT06135558
Title: Presence and Clinical Significance of Marginal Acute Inflammation for Stage II Colon Cancer
Brief Title: Clinical Significance of Marginal Acute Inflammation for Stage II Colon Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, M.D., Sun Yat-sen University
Other Study IDs: GIH-SYip32
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Inflammation; Colon Cancer
MeSH Terms: conditions — Inflammation; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T3: patient staged T3 without marginal acute inflammation
  Interventions: Diagnostic Test: MAI detection
- MAI: patient with marginal acute inflammation
  Interventions: Diagnostic Test: MAI detection
- T4: patient staged T4 without marginal acute inflammation
  Interventions: Diagnostic Test: MAI detection

INTERVENTIONS:
Diagnostic Test: MAI detection — to detect the presence of marginal acute inflammation

SUMMARY:
Marginal acute inflammation would make reporting the serosal involvement of tumors controversial. We aimed to investigate the clinical significance and explore the prognostic value of MAI for stage II localized colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) colon cancer patients with the preoperative staging of stage I-III who lacked distant metastasis; (2) patients who underwent radical resection, with postoperative pathology confirmed as pT3-4N0M0; and (3) complete follow-up information

Exclusion Criteria:

* (1) patients who received neo-adjuvant therapy; (2) patients with multiple primary colorectal cancer; and (3) patients with a history of malignant tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage II colon cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1167 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
DFS | 5 year
  disease free survival

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request